CLINICAL TRIAL: NCT06731140
Title: Reverse HER2-negative Immune Resistant Breast Cancer
Acronym: Resilire
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2411307-7
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-05

CONDITIONS: HER2 Negative Breast Cancer
Keywords: immunotherapy; retinoic acid; HER2 negative breast cancer
MeSH Terms: interventions — Tretinoin; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- retinoic acid with anti-PD-1 immunotherapy (Experimental): retinoic acid with anti-PD-1 immunotherapy
  Interventions: Drug: Retinoic Acid; Drug: anti-PD-1 antibody and chemotherapy

INTERVENTIONS:
Drug: Retinoic Acid — Retinoic acid 20mg tid, p.o.
Drug: anti-PD-1 antibody and chemotherapy — PD-1 antibody SHR1210 200mg q2w chemotherapy (whether and which should be given depends on the treatment regimen before enrollment)

SUMMARY:
This is a Phase II, open-label study evaluating the efficacy and safety of combined treatment (retinoic acid) with immune checkpoint inhibitor in HER2-negative breast cancer patients who progressed during previous immune checkpoint inhibitors.

DETAILED DESCRIPTION:
This is a Phase II, open-label study evaluating the efficacy and safety of combined treatment (retinoic acid) with immune checkpoint inhibitors in metastatic HER2-negative breast cancer patients who progressed during or following previous immune checkpoint inhibitors. HER2-negative breast cancers include luminal breast cancers and triple-negative breast cancers.

Current clinical studies on immunotherapy for luminal breast cancer are limited, with inconsistent results across trials. The KEYNOTE-028 study reported an objective response rate (ORR) of only 12% for pembrolizumab in PD-L1-positive, previously treated advanced luminal breast cancer patients, demonstrating limited efficacy. The GIADA phase II trial revealed a pathological complete response (pCR) rate of 16.3% with neoadjuvant chemotherapy followed by immunotherapy in luminal breast cancer. Additionally, trials such as NCT02779751 and NCT03051659 also indicated limited clinical benefits from immunotherapy. However, the I-SPY2 platform showed that combinations like olaparib, paclitaxel, and immunotherapy or wP-AC chemotherapy with immunotherapy could improve pCR rates in high-risk patients. Despite advancements, immunotherapy benefits are limited in luminal breast cancer compared to other cancers, with advanced-stage patients more likely to develop resistance.

Recent clinical studies on advanced triple-negative breast cancer have shown that immunotherapy combined with chemotherapy demonstrates superior clinical efficacy compared to traditional chemotherapy alone. Phase III trials such as IMPassion130 and Keynote-522 have confirmed that PD-1/PD-L1 inhibitors used with chemotherapy significantly improve progression-free survival, overall survival, and pathological complete response rates. However, compared to other malignancies, triple-negative breast cancer patients still show relatively low overall response rates to immunotherapy: treatment-naïve patients achieve objective response rates of only 10-20% with immunotherapy monotherapy, though this improves to 56% when combined with chemotherapy, extending median progression-free survival to 7.2 months. Unfortunately, efficacy decreases significantly in later treatment lines, with objective response rates falling to just 10.6-15.9% after multiple previous treatments. Thus, strategies to overcome immunotherapy resistance or increase the sensitivity of immunotherapy efficacy are urgently needed for HER2-negative breast cancer patients.

The preclinical results of our center show that retinoic acid can enhance the anti-tumor immune response by promoting the peroxidation of macrophages, increasing the infiltration and function of cytotoxic CD8+ T cells, inhibiting the growth of tumors in mice. Based on the preclinical study, the investigators designed this study to enroll metastatic HER2-negative breast cancer patients who have progressed during or following immunotherapy, and to explore the efficacy of retinoic acid combined with immunotherapy at a clinical level, providing new strategies of combined treatment for HER2-negative breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0, 1, or 2
* Metastatic or locally advanced, histologically confirmed luminal breast cancer (defined as: ER positive when immunohistochemistry shows >1% positive tumor cells, PR positive when >1% tumor cells are positive, and HER2 negative when scored as 0-1+ or when HER2 2+ shows no amplification by FISH or CISH) or triple negative breast cancer (defined as: ER negative when immunohistochemistry shows <1% positive tumor cells, PR negative when <1% tumor cells are positive, and HER2 negative when scored as 0-1+ or when HER2 2+ shows no amplification by FISH or CISH).
* Radiologic/objective evidence of recurrence or disease progression after immunotherapy (combined with targeted therapy or chemo ) for metastatic breast cancer (MBC)
* Adequate hematologic and end-organ function, laboratory test results, obtained within 14 days prior to initiation of study treatment.

For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm

* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* have the cognitive ability to understand the protocol and be willing to participate and to be followed up.

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* Active or history of autoimmune disease or immune deficiency
* Significant cardiovascular disease
* History of malignancy other than breast cancer within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Treatment with chemotherapy, radiotherapy, immunotherapy or surgery (outpatient clinic surgery excluded) within 3 weeks prior to initiation of study treatment.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* History of allergies to the drug components of this trial
* History of eosinophilosis or mastocytosis
* Patients who have been using oral steroid hormones for a long time will need to stop for 4 weeks if they have used them occasionally in the past

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
Clinical Benefit Rate (CBR) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Clinical benefit rate (CBR) is defined as the proportion of subjects who achieve a complete response (CR), partial response (PR), or have durable stable disease (SD) after treatment. It is intended to measure a clinically meaningful and broader disease control effect. CBR includes subjects who have achieved CR and PR, as well as those who have maintained SD for a specified duration (≥24 weeks). The evaluation is based on the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Subjects must have measurable tumor lesions at baseline. The efficacy assessment is categorized into CR, PR, SD, and Progressive Disease (PD) according to RECIST 1.1 criteria.
Immune changes in peripheral blood | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Baseline through end of study, assessed up to 6 months
Progression Free Survival (PFS) | Randomization to death from any cause, through the end of study, assessed up to 6 months
Safety and treatment-related AEs | Randomization to death from any cause, through the end of study, assessed up to 12 months
Biomarker analysis | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Retinoic acid related genes, cell functions and microbes will be measured in pre-treatment and post-treatment samples (tumor tissue, blood and fecal samples) to predict therapy response.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided